CLINICAL TRIAL: NCT05413642
Title: Prevention of Hospitalization of Patients With Early COVID-19 by an Anti-inflammatory Drug-based Home-treatment Algorithm:a Three-months, Pragmatic, Cluster Randomized, Open-label, Blinded Endpoint (PROBE) Trial
Brief Title: COVID-19 Algorithm Treatment at Home
Acronym: COVER-HOME
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to changes in the monitoring rules for SARS-CoV-2 and the dramatic reduction in COVID-19 cases, it became extremely difficult to recruit the required number of patients provided by the study protocol to meet the study's primary objective.
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVER-HOME; 2022-001474-64 (EudraCT Number)
Record Dates: First submitted 2022-06-09; First posted 2022-06-10 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: COVID-19 treatment at home; Early symptoms; Hospitalization; Anti-inflammatory drugs
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Recommended algorithm' cohort (Experimental): COVID-19 patients treated at home by their family doctors according to the proposed recommendations
  Interventions: Drug: Recommended treatment schedule
- Usual care (Active Comparator): COVID-19 patients treated at home by their family doctors according to their usual clinical practice expected to be in accordance with AIFA recommendations
  Interventions: Drug: Usual care

INTERVENTIONS:
Drug: Recommended treatment schedule — Non-steroidal anti-inflammatory drugs (NSAIDs) Corticosteroids (Dexamethasone), Anticoagulants (LMW heparin), Gentle oxygen therapy
  Arms: 'Recommended algorithm' cohort
Drug: Usual care — Treatment regimens different from the recommended one according to family physician personal practice
  Arms: Usual care

SUMMARY:
The newly recognised disease COVID-19 is caused by the Severe-Acute-Respiratory-Syndrome Coronavirus 2 (SARS-CoV-2), which rapidly spread globally in late 2019, reaching pandemic proportions. The clinical spectrum of SARS-CoV-2 infection is broad, encompassing asymptomatic infection, mild upper respiratory tract illness and mild extrapulmonary symptoms, and severe viral pneumonia with respiratory failure and even death.

For COVID-19, most primary care physicians have initially treated their patients at home according to their judgment, with various treatment regimens they believe are most appropriate based on their experience/expertise. We recently published a note on how we were treating patients at home based on the pathophysiology underlining the mild/moderate symptoms at the onset of the illness and the proposal of simple drugs that theoretically better fit these mechanisms.

Because the common early mild symptoms of COVID-19 highlight a systemic inflammatory process, there is the recommendation of using anti-inflammatory agents to limit excessive host inflammatory responses to the viral infection, including non-steroidal anti-inflammatory drugs and corticosteroids. Moreover, COVID-19 patients are exposed to the risk of thromboembolic events and anticoagulant prophylaxis is recommended even at home, in particular settings, unless contraindicated.

In an academic matched-cohort study, we found that early treatment of COVID-19 patients at home by their family doctors according to the proposed recommendation regimen almost completely prevented the need for hospital admission (the most clinically relevant outcome of the study along with death) due to progression toward more severe illness (2 out of 90 patients), compared to patients in the 'control' cohort who were treated at home according to their family physician's assessments (13 out of 90 patients). However, the rate of hospitalization was a secondary outcome of the study and the possibility of a casual finding cannot be definitely excluded. Moreover, these findings were achieved in a retrospective observational study with two matched cohorts of COVID-19 patients, a possible additional limitation of the robustness of the conclusions that would deserve further validation. Thus, we have considered the observed reduction in patient hospitalization a hypothesis generating finding to be confirmed.

In this pragmatic, prospective, three-months, cluster randomized, open-label, blinded endpoint (PROBE) clinical trial, we will compare two groups of family doctors according to a randomized approach, who will treat their COVID19-patients with the proposed recommendation algorithm or other treatment regimens they normally feel appropriate according to their usual clinical practice, and monitor them longitudinally up to 3 months.

Our working hypothesis is that following the proposed recommendation algorithm the early COVID-19-related inflammatory process is limited, preventing the need of hospital admission at larger extent than with other therapeutic approaches also targeting early symptoms of the illness at home.

Should the findings be confirmed, the tested standardized treatment protocol would achieve major benefits for patients with early COVID-19 in particular in relation to a remarkably reduced risk of hospitalization that is expected to translate into reduced morbility and, possibly, mortality. Notably, these expected clinical benefits would be associated with remarkably reduced treatment costs related to reduced hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult (≥18 years old)
* Subjects with early mild/moderate symptoms of COVID-19*, who start the treatment without waiting results of a nasopharyngeal swab**

  * Influenza-like syndrome, (i.e. flu, cough, myalgias/arthralgias or other painful symptoms, fever, gastrointestinal symptoms), no dyspnea, SpO2 >94%, or asthenia,ageusia/dysgeusia, anosmia, or MEWS 0 to 3.

  ** Nasopharyngeal swab should be performed soon after the onset of symptoms possibly related to SARS-CoV-2
* Subjects without known comorbidities in their previous medical history
* Subjects with known comorbidities that bring them at high risk of COVID-19 progression (heart disease, hypertension, asthma or lung disease, diabetes, chronic kidney disease, stroke or neurological problems, weakened immune system - e.g. receiving chemotherapy -, and self-reported obesity or body-mass index of at least 30 kg/sqm)
* Informed consent

Exclusion Criteria:

* Subjects who require immediate hospital admission because of severe COVID-19 symptoms at onset according to family doctor's assessment (MEWS score 5, and/or septic shock, multiorgan failure)
* Known hypersensitivity or allergy to any medication under investigation
* Specific contraindications to the use of each recommended drugs according to their summary of product characteristics and the clinical judgment of family doctor
* Legal incapacity, limited legal incapacity, intellectual disability, uncooperative attitude or any other evidence that the patient will not be able to understand the study aims and procedures
* Pregnancy* (*Patient with childbearing potential will be included according to the pragmatic design of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
proportion of patients who reach score ≥ 5 of MEWS, an index of the need of hospitalization, in the two treatment groups | From beginning the proposed recommended treatments or other therapeutic regimens, assessed up to 90 days)